CLINICAL TRIAL: NCT02244463
Title: A Phase I/II Study of MLN0128 in Metastatic Anaplastic Thyroid Cancer and Incurably Poorly Differentiated or Radioidodine Refractory Differentiated Thyroid Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Kartik Sehgal, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-223
Record Dates: First submitted 2014-09-17; First posted 2014-09-19 (Estimated); Results first posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2023-12

CONDITIONS: Anaplastic Thyroid Cancer; Thyroid Cancer; Differentiated Thyroid Cancer
Keywords: Anaplastic Thyroid Cancer; Thyroid Cancer; Differentiated Thyroid Cancer
MeSH Terms: conditions — Thyroid Carcinoma, Anaplastic; Thyroid Neoplasms | interventions — sapanisertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Phase I: Dose Level 1 (PI DL1) (Experimental): Phase I Dose Level 1 participants receive MLN0128 3 mg orally, daily for 28 days. Participants are treated until disease progression or withdrawal of consent.
  Interventions: Drug: MLN0128
- Phase I: Dose Level 2 (PI DL2) (Experimental): Phase I Dose Level 3 (dose escalation) participants received MLN0128 5 mg orally, daily for 28 days. Participants are treated until disease progression or withdrawal of consent.
  Interventions: Drug: MLN0128
- Phase I: Dose Level 3 (PI DL3) (Experimental): Phase I Dose Level 3 participants receive MLN0128 5 mg orally, daily for 28 days. Participants are treated until disease progression or withdrawal of consent.
  Interventions: Drug: MLN0128
- Phase I: Dose Level 3 (PI DL3) Expansion (Experimental): Phase I Dose Level 3 participants receive MLN0128 5 mg orally, daily for 28 days. Participants are treated until disease progression or withdrawal of consent.
  Interventions: Drug: MLN0128
- Phase II: ATC Cohort (Experimental): Phase II participants receive MLN0128 at the recommended phase II dose of 5 mg orally, daily for 28 days. Participants are treated until disease progression or withdrawal of consent. All phase I participants treated at the maximum tolerated dose/ recommended phase II dose (DL3) are enrolled in the phase II part of the study according to the appropriate disease cohort.
  Interventions: Drug: MLN0128
- Phase II: DTC Cohort (Experimental): Phase II participants receive MLN0128 at the recommended phase II dose of 5 mg orally, daily for 28 days. Participants are treated until disease progression or withdrawal of consent. All phase I participants treated at the maximum tolerated dose/ recommended phase II dose (DL3) are enrolled in the phase II part of the study according to the appropriate disease cohort.
  Interventions: Drug: MLN0128

INTERVENTIONS:
Drug: MLN0128
  Other Names: INK128; Sapanisertib

SUMMARY:
This research study is a phase I/II study of MLN0128 in metastatic anaplastic thyroid cancer(ATC) and incurably poorly differentiated or radioidodine refractory differentiated thyroid cancer (DTC).

Due to changes in the manufacturing process which resulted in increased absorption of MLN0128 from capsules, a run-in phase I prior to the phase II of the study was needed.

Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied. The FDA (the U.S. Food and Drug Administration) has not approved MLN0128 as a treatment for any disease.

MLN0128 prevents tumor cells from dividing and growing by selectively and potently inhibiting a chemical, mTOR kinase, which regulates cell growth and survival. Patients with anaplastic thyroid cancer have been observed to sometimes carry genetic alterations in their tumor cells which may make the cancer more sensitive to inhibition by MLN0128.

Given the activity with everolimus in RAI refractory thyroid cancer, subjects wth metastatic, incurable differentiated RAI refractory and poorly differentiated thyroid cancer were included.

DETAILED DESCRIPTION:
Patients who fulfill eligibility criteria will be entered into the trial to receive MLN0128.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years or older
* Any number of prior chemotherapy or targeted agents including rapamycin analogues allowed
* Newly diagnosed or refractory/metastatic anaplastic thyroid cancer confirmed by histology, incurable by surgery, radiotherapy or chemoradiotherapy alone or in combination
* Must have measurable disease
* ECOG performance status 0-2
* No active intracranial metastases
* Tissue for correlative studies must be available
* Ability to swallow oral medications
* Voluntary written consent must be given before performance of any study related procedure
* Adequate organ function, as specified below, within 21 days:

  * Bone marrow reserve consistent with: absolute neutrophil count (ANC) ≥ 1.5 x 109/L; platelet count ≥ 100 x 109/L; hemoglobin ≥ 9 g/dL;
  * Hepatic: total bilirubin ≤1.5 x upper limit of normal (ULN), transaminases (aspartate aminotransferase/serum glutamic oxaloacetic transaminase-AST/SGOT and alanine aminotransferase/serum glutamic pyruvic transaminase-ALT/SGPT) ≤2.5 x ULN (≤5 x ULN if liver metastases are present);
  * Renal: creatinine clearance ≥50 mL/min
  * Metabolic: fasting serum glucose (≤ 130 mg/dL) and fasting triglycerides ≤ 300 mg/dL
  * Left ventricular ejection fraction (LVEF) within 5 absolute percentage points of institutional standard of normal as measured by echocardiogram (ECHO) or multiple gated acquisition scan (MUGA) within 4 weeks prior to first study drug administration (ie, if the institutional normal is 50%, subject's LVEF may be as low as 45% to be eligible for the study)
* Female patients who:

  * Are postmenopausal for at least 1 year before the screening visit, OR
  * Are surgically sterile, OR
  * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 90 days after the last dose of study drug, or agree to completely abstain from heterosexual intercourse
* Male patients, even if surgically sterilized (ie, status post-vasectomy), who:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, or
  * Agree to completely abstain from heterosexual intercourse
* Treatment with strong CYP2C19, CYP3A4, and CYP2C9 inhibitors and/or inducers must be discontinued

Exclusion Criteria:

* Female patients who are both lactating and breastfeeding or have a positive serum pregnancy test during the screening period
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment
* Treatment with any investigational products within 14 days
* Failed to recover from the reversible effects of prior anticancer therapies
* Manifestations of malabsorption due to prior gastrointestinal surgery or disease
* Poorly controlled diabetes mellitus
* History of any of the following within the last 6 months prior to study entry:

  * Ischemic myocardial event
  * Ischemic cerebrovascular event
  * Requirement for inotropic support (excluding digoxin) or serious (uncontrolled) cardiac arrhythmia
  * Placement of a pacemaker for control of rhythm
  * New York Heart Association Class III or IV heart failure
  * Pulmonary embolism
* Significant active cardiovascular or pulmonary disease at the time of study entry, including:

  * Uncontrolled high blood pressure
  * Pulmonary hypertension
  * Uncontrolled asthma or O2 saturation < 90%
  * Significant valvular disease
  * Medically significant (symptomatic) bradycardia
  * History of arrhythmia requiring an implantable cardiac defibrillator
  * Baseline prolongation of the rate-corrected QT interval (QTc)
* Treatment with hematopoietic growth factors, transfusions of blood and blood products, or systemic corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kartik Seghal, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Medical School, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data. Cumulative results will be posted here and published.

REFERENCES:
- [Derived] Cabanillas ME, McFadden DG, Durante C. Thyroid cancer. Lancet. 2016 Dec 3;388(10061):2783-2795. doi: 10.1016/S0140-6736(16)30172-6. Epub 2016 May 27. PMID 27240885

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled from July 2015 to July 2020.
Groups:
- Phase I: Dose Level 1 (PI: DL1): Phase I Dose Level 1 participants received MLN0128 3 mg orally, daily for 28 days. Participants are treated until disease progression or withdrawal of consent.
- Phase I: Dose Level 2 (PI: DL2): Phase I Dose Level 2 participants received MLN0128 4 mg orally, daily for 28 days. Participants are treated until disease progression or withdrawal of consent.
- Phase I: Dose Level 3 (PI: DL3): Phase I Dose Level 3 (dose escalation) participants received MLN0128 5 mg orally, daily for 28 days. Participants are treated until disease progression or withdrawal of consent.
- Phase I: Dose Level 3 Expansion (PI: DL3 Exp): Phase 1 Dose Level 3 participants receive MLN0128 5 mg orally, daily for 28 days. Participants are treated until disease progression or withdrawal of consent.
- Phase II: ATC Cohort; Phase II: DTC Cohort: Phase II participants receive MLN0128 at the recommended phase II dose of 5 mg orally, daily for 28 days. Participants are treated until disease progression or withdrawal of consent. All phase I participants treated at the maximum tolerated dose/ recommended phase II dose (DL3) were also enrolled in the phase II part of the study according to the appropriate disease cohort.
Period: Period 1: PI DL1 Dose Escalation
Arm/Group | Phase I: Dose Level 1 (PI: DL1) | Phase I: Dose Level 2 (PI: DL2) | Phase I: Dose Level 3 (PI: DL3) | Phase I: Dose Level 3 Expansion (PI: DL3 Exp) | Phase II: ATC Cohort | Phase II: DTC Cohort
Started | 3 | 0 | 0 | 0 | 0 | 0
Completed (Given treatment duration is not fixed, all participants are considered as 'Non Completed' and reason off-treatment provided.) | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Disease Progression | 3 | 0 | 0 | 0 | 0 | 0
Period: Period 2: PI DL2 Dose Escalation
Arm/Group | Phase I: Dose Level 1 (PI: DL1) | Phase I: Dose Level 2 (PI: DL2) | Phase I: Dose Level 3 (PI: DL3) | Phase I: Dose Level 3 Expansion (PI: DL3 Exp) | Phase II: ATC Cohort | Phase II: DTC Cohort
Started (The 'NOTE' here is an error: Each subsequent period in the PI study involves new participants.) | 0 | 3 | 0 | 0 | 0 | 0
Completed (Given treatment duration is not fixed, all participants are considered as 'Non Completed' and reason off-treatment provided.) | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Disease Progression | 0 | 2 | 0 | 0 | 0 | 0
Period: Period 3: PI DL3 Dose Escalation
Arm/Group | Phase I: Dose Level 1 (PI: DL1) | Phase I: Dose Level 2 (PI: DL2) | Phase I: Dose Level 3 (PI: DL3) | Phase I: Dose Level 3 Expansion (PI: DL3 Exp) | Phase II: ATC Cohort | Phase II: DTC Cohort
Started (The 'NOTE' here is an error: Each subsequent period in the PI study involves new participants.) | 0 | 0 | 3 | 0 | 0 | 0
Completed (Given treatment duration is not fixed, all participants are considered as 'Non Completed' and reason off-treatment provided.) | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 3 | 0 | 0 | 0
Not completed — Disease Progression | 0 | 0 | 3 | 0 | 0 | 0
Period: Period 4: PI DL3 Dose Expansion
Arm/Group | Phase I: Dose Level 1 (PI: DL1) | Phase I: Dose Level 2 (PI: DL2) | Phase I: Dose Level 3 (PI: DL3) | Phase I: Dose Level 3 Expansion (PI: DL3 Exp) | Phase II: ATC Cohort | Phase II: DTC Cohort
Started (The 'NOTE' here is an error: Each subsequent period in the PI study involves new participants.) | 0 | 0 | 0 | 10 | 0 | 0
Completed (Given treatment duration is not fixed, all participants are considered as 'Non Completed' and reason off-treatment provided.) | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 10 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Disease Progression | 0 | 0 | 0 | 5 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Intercurrent Illness | 0 | 0 | 0 | 1 | 0 | 0
Period: Period 5: Phase II
Arm/Group | Phase I: Dose Level 1 (PI: DL1) | Phase I: Dose Level 2 (PI: DL2) | Phase I: Dose Level 3 (PI: DL3) | Phase I: Dose Level 3 Expansion (PI: DL3 Exp) | Phase II: ATC Cohort | Phase II: DTC Cohort
Started (The 'NOTE' here is an error: the PII study total sample size is unrelated to the previous PI study. Per design, all participants treated at the maximum tolerated dose would be enrolled in the PII study. In the ATC and DTC PII cohorts, there were n=6 and n=7 participants, respectively, who received the RP2D in the PI study (DL3 escalation and expansion). There were n=12 (ATC) and n=15 (DTC) participants who subsequently enrolled in the PII study.) | 0 | 0 | 0 | 0 | 18 | 22
Completed (Given treatment duration is not fixed, all participants are considered as 'Non Completed' and reason off-treatment provided.) | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 18 | 22
Not completed — Disease Progression | 0 | 0 | 0 | 0 | 10 | 11
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 3 | 4
Not completed — Intercurrent Illness | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Still On treatment | 0 | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of all enrolled participants.
Groups:
- P1: DL1: Phase I Dose Level 1 participants received MLN0128 3 mg orally, daily for 28 days. Participants are treated until disease progression or withdrawal of consent.
- PI: DL2: Phase I Dose Level 2 participants received MLN0128 4 mg orally, daily for 28 days. Participants are treated until disease progression or withdrawal of consent.
- PI: DL3: Phase I Dose Level 3 (dose escalation) participants received MLN0128 5 mg orally, daily for 28 days. Participants are treated until disease progression or withdrawal of consent.
- P1: DL3 EXP: Phase 1 Dose Level 3 participants receive MLN0128 5 mg orally, daily for 28 days. Participants are treated until disease progression or withdrawal of consent.
- Phase II: ATC Cohort (Including DL3 PI); Phase II: DTC Cohort (Including DL3 PI): Phase II participants receive MLN0128 at the maximum tolerated dose/ recommended phase II dose of 5 mg orally, daily for 28 days. Participants are treated until disease progression or withdrawal of consent. Per design, all participants treated at the maximum tolerated dose (DL3) would be enrolled in the PII study.
- Total: Total of all reporting groups
Arm/Group | P1: DL1 | PI: DL2 | PI: DL3 | P1: DL3 EXP | Phase II: ATC Cohort (Including DL3 PI) | Phase II: DTC Cohort (Including DL3 PI) | Total
Number analyzed (Participants) | 3 | 3 | 3 | 10 | 18 | 22 | 59
Age, Continuous [Median (Full Range); unit: years] — Population: Per design, all participants treated at the maximum tolerated dose (DL3) would be enrolled in the PII study and, as such, these participants are included for both PI and PII representation. PII data include n=6 ATC participants and n=7 DTC participants from the PI study.
  years
    Phase I: number analyzed (Participants) | 3 | 3 | 3 | 10 | 0 | 0 | 19
    Phase I | 59.3 [53.9 to 74.4] | 75.8 [69.5 to 77.6] | 55.7 [51.5 to 82.4] | 65.7 [50.7 to 86.2] |  |  | 67.7 [50.7 to 86.2]
    Phase II: number analyzed (Participants) | 0 | 0 | 0 | 0 | 18 | 22 | 40
    Phase II |  |  |  |  | 64.6 [52.5 to 86.2] | 66.2 [37.9 to 86.5] | 65.5 [37.9 to 86.5]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Per design, all participants treated at the maximum tolerated dose (DL3) would be enrolled in the PII study and, as such, these participants are included for both PI and PII representation. PII data include n=6 ATC participants and n=7 DTC participants from the PI study.
  Participants
    Phase I: number analyzed (Participants) | 3 | 3 | 3 | 10 | 0 | 0 | 19
    Phase I: Female | 2 | 1 | 1 | 5 |  |  | 9
    Phase I: Male | 1 | 2 | 2 | 5 |  |  | 10
    Phase II: number analyzed (Participants) | 0 | 0 | 0 | 0 | 18 | 22 | 40
    Phase II: Female |  |  |  |  | 11 | 11 | 22
    Phase II: Male |  |  |  |  | 7 | 11 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Per design, all participants treated at the maximum tolerated dose (DL3) would be enrolled in the PII study and, as such, these participants are included for both PI and PII representation. PII data include n=6 ATC participants and n=7 DTC participants from the PI study.
  Participants
    Phase I: number analyzed (Participants) | 3 | 3 | 3 | 10 | 0 | 0 | 19
    Phase I: Hispanic or Latino | 0 | 1 | 0 | 0 |  |  | 1
    Phase I: Not Hispanic or Latino | 3 | 2 | 3 | 10 |  |  | 18
    Phase I: Unknown or Not Reported | 0 | 0 | 0 | 0 |  |  | 0
    Phase II: number analyzed (Participants) | 0 | 0 | 0 | 0 | 18 | 22 | 40
    Phase II: Hispanic or Latino |  |  |  |  | 0 | 1 | 1
    Phase II: Not Hispanic or Latino |  |  |  |  | 18 | 21 | 39
    Phase II: Unknown or Not Reported |  |  |  |  | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Per design, all participants treated at the maximum tolerated dose (DL3) would be enrolled in the PII study and, as such, these participants are included for both PI and PII representation. PII data include n=6 ATC participants and n=7 DTC participants from the PI study.
  Participants
    Phase I: number analyzed (Participants) | 3 | 3 | 3 | 10 | 0 | 0 | 19
    Phase I: White | 3 | 2 | 3 | 10 |  |  | 18
    Phase I: Black/African American | 0 | 0 | 0 | 0 |  |  | 0
    Phase I: Other | 0 | 1 | 0 | 0 |  |  | 1
    Phase II: number analyzed (Participants) | 0 | 0 | 0 | 0 | 18 | 22 | 40
    Phase II: White |  |  |  |  | 17 | 21 | 38
    Phase II: Black/African American |  |  |  |  | 1 | 0 | 1
    Phase II: Other |  |  |  |  | 0 | 1 | 1
Eastern Cooperative Oncology Group Performance Score (ECOG PS) [Count of Participants; unit: Participants] — ECOG PS0: Fully active, able to carry on all pre-disease performance without restriction ECOG PS1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature ECOG PS2: Ambulatory and capable of all self-care but unable to carry out any work activities; Up and about more than 50% of waking hours Population: Per design, all participants treated at the maximum tolerated dose (DL3) would be enrolled in the PII study and, as such, these participants are included for both PI and PII representation. PII data include n=6 ATC participants and n=7 DTC participants from the PI study.
  Participants
    Phase I: number analyzed (Participants) | 3 | 3 | 3 | 10 | 0 | 0 | 19
    Phase I: ECOG PS0 | 0 | 1 | 0 | 3 |  |  | 4
    Phase I: ECOG PS1 | 2 | 2 | 3 | 7 |  |  | 14
    Phase I: ECOG PS2 | 1 | 0 | 0 | 0 |  |  | 1
    Phase II: number analyzed (Participants) | 0 | 0 | 0 | 0 | 18 | 22 | 40
    Phase II: ECOG PS0 |  |  |  |  | 5 | 0 | 5
    Phase II: ECOG PS1 |  |  |  |  | 12 | 21 | 33
    Phase II: ECOG PS2 |  |  |  |  | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) [Phase I Dose Escalation]
Description: The MTD is determined by the number of participants who experience a dose limiting toxicity (DLT). The MTD is defined as the highest dose at which fewer than one-third of participants experience a DLT. If no DLTs are observed, the MTD is not reached but the highest dose received may be the Recommended Phase II Dose (RP2D).
Time Frame: cycle 1 (cycle duration=28 days)
Population: The analysis datasets reflects participants who enrolled on the phase I dose escalation study.
Measure: Number; unit: mg
Groups:
- All Phase I Dose Escalation Participants: All phase I dose escalation participants receive MLN0128 orally, daily for 28 days according to the dose escalation schedule. Participants are treated until disease progression or withdrawal of consent.
Arm/Group | All Phase I Dose Escalation Participants
Number analyzed (Participants) | 9
mg | 5

2. Primary Outcome: Number of Participants With Dose Limiting Toxicity (DLT) [Phase I Dose Escalation]
Description: DLT is defined as an adverse event based on the Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0) or abnormal laboratory value assessed as unrelated to disease, disease progression, intercurrent illness, or concomitant medications, that meets any of the criteria (hematologic, renal, hepatic, endocrine, metabolic/laboratory, pancreatitis, cardiac, neurotoxicity, mood alteration, dermatologic] listed in section 5.3.2 of the protocol.
Time Frame: cycle 1 (cycle duration=28 days)
Population: The analysis population is comprised of all participants enrolled in the PI dose escalation design.
Measure: Count of Participants; unit: Participants
Groups:
- Phase I: Dose Level 2 (PI DL2): Phase I Dose Level 2 participants receive MLN0128 4 mg orally, daily for 28 days. Participants are treated until disease progression or withdrawal of consent.
Arm/Group | Phase I: Dose Level 1 (PI DL1) | Phase I: Dose Level 2 (PI DL2) | Phase I: Dose Level 3 (PI DL3)
Number analyzed (Participants) | 3 | 3 | 3
Participants | 0 | 0 | 0

3. Primary Outcome: 4-month Progression Free Survival (PFS4) Rate - ATC Cohort [Phase II]
Description: PFS4 rate is the percentage of participants remaining alive and progression-free at 4-months from study entry. Per RECIST 1.1 for target lesions: disease progression (PD) is at least a 20% increase in sum longest diameter (LD), taking as reference the smallest sum on study with at least 5 mm absolute increase or the appearance of one or more new lesions. For non-target lesions, PD is appearance of one or more new lesions or unequivocal progression of existing non-target lesions.
Time Frame: Disease was assessed radiologically every 2 cycles/ 8 weeks on treatment until the earliest of first progression, death or 24 months from study entry. Relevant for this endpoint was observation at 4-months.
Population: The analysis dataset is comprised of all participants enrolled to the Phase II ATC cohort.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II: ATC Cohort
Number analyzed (Participants) | 18
percentage of participants | 11.1 [2.0 to 31.0]

4. Secondary Outcome: Number of Participants With Grade 3-5 Treatment-related Toxicity [Phase I/Phase II]
Description: All grade 3-5 adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv4 as reported on case report forms were counted. Maximum grade toxicity by AE type was then calculated. Incidence is the number of participants experiencing at least one grade 2-5 treatment-related AE during the time of observation.
Time Frame: Assessed on treatment at cycles 1 and 2 (days 1 and 15), cycle 3+ on day 1, at the end of treatment and up to 30 days post-treatment. Participants were on treatment up to 21.6 months (median 2.1 months).
Population: The analysis dataset is comprised of all participants enrolled to the study.
Measure: Count of Participants; unit: Participants
Groups:
- PI DL1: Phase I Dose Level 1 participants received MLN0128 3 mg orally, daily for 28 days. Participants are treated until disease progression or withdrawal of consent.
- PI DL2: Phase I Dose Level 2 participants received MLN0128 4 mg orally, daily for 28 days. Participants are treated until disease progression or withdrawal of consent.
- PI DL3: Phase I Dose Level 3 (dose escalation) participants received MLN0128 5 mg orally, daily for 28 days. Participants are treated until disease progression or withdrawal of consent.
- PI DL3 Exp: Phase 1 Dose Level 3 participants receive MLN0128 5 mg orally, daily for 28 days. Participants are treated until disease progression or withdrawal of consent.
Arm/Group | PI DL1 | PI DL2 | PI DL3 | PI DL3 Exp | Phase II: ATC Cohort | Phase II: DTC Cohort
Number analyzed (Participants) | 3 | 3 | 3 | 10 | 18 | 22
Participants | 0 | 1 | 0 | 3 | 4 | 8

5. Secondary Outcome: 6-month Progression Free Survival (PFS6) Rate - DTC Cohort [Phase II]
Description: PFS6 rate is the percentage of patients remaining alive and progression-free at 6-months from study entry. Per RECIST 1.1 for target lesions: disease progression (PD) is at least a 20% increase in sum longest diameter (LD), taking as reference the smallest sum on study with at least 5 mm absolute increase or the appearance of one or more new lesions. For non-target lesions, PD is appearance of one or more new lesions or unequivocal progression of existing non-target lesions.
Time Frame: Disease was assessed radiologically every 2 cycles/ 8 weeks on treatment until the earliest of first progression, death or 24 months from study entry. Relevant for this endpoint was observation at 6-months.
Population: The analysis dataset is comprised of all participants enrolled to the Phase II DTC cohort.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II: DTC Cohort
Number analyzed (Participants) | 22
percentage of participants | 45.5 [27.1 to 64.7]

6. Secondary Outcome: Overall Response Rate (ORR) [Phase II]
Description: ORR was defined as the percentage of participants achieving complete response (CR) or partial response (PR) based on RECIST 1.1 criteria. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions; PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. Confirmatory scan obtained 8 weeks following initial documentation of objective response.
Time Frame: Disease was assessed radiologically every 2 cycles/ 8 weeks on treatment until the earliest of first progression, death or 24 months from study entry. Participants were on treatment up to 196 days (PII ATC) and 454 days (PII DTC).
Population: The analysis dataset is comprised of all participants enrolled to the Phase II ATC and DTC cohorts.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II: ATC Cohort | Phase II: DTC Cohort
Number analyzed (Participants) | 18 | 22
percentage of participants | 0 [0 to 15.3] | 1 [0.2 to 19.8]

7. Secondary Outcome: Median Overall Survival (OS) [Phase II]
Description: OS based on the Kaplan-Meier method is defined as the time from study entry to death or censored at date last known alive.
Time Frame: Long term follow-up for survival was every 3 months post-treatment end up to 24 months.
Population: The analysis dataset is comprised of all participants enrolled to the Phase II ATC and DTC cohorts.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II: ATC Cohort | Phase II: DTC Cohort
Number analyzed (Participants) | 18 | 22
months | 6.1 [4 to 10.3] | 20.4 [17.3 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants had experienced an event (death) as of the final analysis.

8. Secondary Outcome: BRAF V600E Status [Phase II]
Description: Participants were classified by BRAF V600E mutation status evaluated by next generation sequencing (NGS) platforms using tumor tissue collected at baseline.
Time Frame: Baseline
Population: The analysis dataset is comprised of participants with evaluable baseline samples.
Measure: Count of Participants; unit: Participants
Groups:
- Phase II: ATC Cohort; Phase II: DTC Cohort: Phase II participants receive MLN0128 at the maximum tolerated dose/ recommended phase II dose of 5 mg orally, daily for 28 days. Participants are treated until disease progression or withdrawal of consent. Per design, all participants treated at the maximum tolerated dose (DL3) would be enrolled in the PII study.
Arm/Group | Phase II: ATC Cohort | Phase II: DTC Cohort
Number analyzed (Participants) | 11 | 16
Participants
  Absent | 7 | 8
  Present | 4 | 8

9. Secondary Outcome: Clinical Benefit (CBR) by BRAF V600E Status [Phase II]
Description: CBR was defined as the percentage of participants achieving complete response (CR), partial response (PR) or stable disease (SD) based on RECIST 1.1 criteria. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions; PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. Confirmatory scan obtained 8 weeks following initial documentation of CR or PR. SD is neither PR or better nor PD (defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum since treatment start, or the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions). Participants were classified by BRAF V600E status based on established methods using tumor tissue collected at baseline.
Time Frame: BRAF V600E status per NGS at baseline. Disease response was assessed every 2 cycles on treatment until the first progression, death or 24 months from study entry. Participants were on treatment up to 196 days (PII ATC) and 454 days (PII DTC).
Population: The analysis dataset is comprised of participants with evaluable baseline samples.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Phase II: ATC Cohort BRAF V600E Present; Phase II: ATC Cohort BRAF V600E Absent; Phase II: DTC Cohort BRAF V600E Present Status; Phase II: DTC Cohort BRAF V600E Absent Status: Phase II participants receive MLN0128 at the recommended phase II dose of 5 mg orally, daily for 28 days. Participants are treated until disease progression or withdrawal of consent. All phase I participants treated at the maximum tolerated dose/ recommended phase II dose (DL3) were also enrolled in the phase II part of the study according to the appropriate disease cohort. BRAF V600E status was determined at baseline.
Arm/Group | Phase II: ATC Cohort BRAF V600E Present | Phase II: ATC Cohort BRAF V600E Absent | Phase II: DTC Cohort BRAF V600E Present Status | Phase II: DTC Cohort BRAF V600E Absent Status
Number analyzed (Participants) | 4 | 7 | 8 | 8
percentage of participants | 25 [1 to 75] | 28.6 [5 to 66] | 87.5 [53 to 99] | 75.0 [40 to 95]

ADVERSE EVENTS:
Time Frame: Assessed on treatment at cycles 1 and 2 (days 1 and 15), cycle 3+ on day 1, at the end of treatment and up to 30 days post-treatment. Participants were on treatment up to 21.6 months (median 2.1 months).
Description: Serious AEs (SAE) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher. All remaining AEs are classified as Other AEs (OAE) including grade 3 or higher events with treatment-attribution of unlikely and unrelated plus all grade 1 and 2 events. Maximum grade toxicity by type was then calculated within SAE and OAE datasets. No further data is available to specify classification of other beyond the general term.
Groups:
- PI: DL1: Phase I: DL1 participants receive MLN0128 3 mg orally, daily for 28 days according to the dose escalation schedule. Participants are treated until disease progression or withdrawal of consent.
- PI: DL2: Phase I: DL2 participants receive MLN0128 4mg orally, daily for 28 days according to the dose escalation schedule. Participants are treated until disease progression or withdrawal of consent.
- PI: DL3 Exp: Phase 1 Dose Level 3 participants receive MLN0128 5 mg orally, daily for 28 days. Participants are treated until disease progression or withdrawal of consent.
- Phase II: ATC Cohort (Including P1 DL3); Phase II: DTC Cohort (Including P1 DL3): Phase II participants receive MLN0128 at the recommended phase II dose of 5 mg orally, daily for 28 days. Participants are treated until disease progression or withdrawal of consent. All phase I participants treated at the maximum tolerated dose/ recommended phase II dose (DL3) were also enrolled in the phase II part of the study according to the appropriate disease cohort.
Arm/Group | PI: DL1 | PI: DL2 | PI: DL3 | PI: DL3 Exp | Phase II: ATC Cohort | Phase II: DTC Cohort | Phase II: ATC Cohort (Including P1 DL3) | Phase II: DTC Cohort (Including P1 DL3)
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/3 | 0/3 | 0/10 | 0/12 | 0/15 | 0/18 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 0/3 | 3/10 | 3/12 | 6/15 | 4/18 | 8/22
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 10/10 | 12/12 | 15/15 | 18/18 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PI: DL1 (N=3) | PI: DL2 (N=3) | PI: DL3 (N=3) | PI: DL3 Exp (N=10) | Phase II: ATC Cohort (N=12) | Phase II: DTC Cohort (N=15) | Phase II: ATC Cohort (Including P1 DL3) (N=18) | Phase II: DTC Cohort (Including P1 DL3) (N=22)
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 3
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PI: DL1 (N=3) | PI: DL2 (N=3) | PI: DL3 (N=3) | PI: DL3 Exp (N=10) | Phase II: ATC Cohort (N=12) | Phase II: DTC Cohort (N=15) | Phase II: ATC Cohort (Including P1 DL3) (N=18) | Phase II: DTC Cohort (Including P1 DL3) (N=22)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 3 | 0 | 2 | 1 | 5
Alkaline phosphatase increased (Investigations) | 1 | 0 | 1 | 1 | 1 | 2 | 2 | 3
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 1
Anorexia (Metabolism and nutrition disorders) | 3 | 2 | 0 | 5 | 6 | 8 | 8 | 11
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 4 | 2 | 5 | 2 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 2 | 3 | 1 | 2 | 2 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 4 | 3 | 4 | 3
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Blurred vision (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain - cardiac (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Chills (General disorders) | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 3
Cholesterol high (Investigations) | 0 | 0 | 0 | 1 | 4 | 8 | 4 | 9
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Confusion (Psychiatric disorders) | 1 | 1 | 0 | 1 | 1 | 1 | 2 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 2 | 2 | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1 | 5 | 5 | 3 | 9 | 5
Creatinine increased (Investigations) | 0 | 0 | 2 | 3 | 1 | 3 | 4 | 5
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 1 | 2 | 2 | 1 | 3 | 3
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 2 | 3 | 2 | 4
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0 | 6 | 4 | 11 | 8 | 13
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 2 | 3 | 6 | 5 | 7
Dry eye (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 1 | 2 | 3 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 3 | 1 | 2 | 2 | 4
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 1 | 1 | 2 | 2 | 2
Dysphagia (Gastrointestinal disorders) | 2 | 1 | 0 | 2 | 4 | 4 | 6 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 3 | 2 | 8 | 4 | 11
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1
Edema face (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1
Edema limbs (General disorders) | 1 | 0 | 2 | 4 | 1 | 3 | 3 | 7
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 2
Endocrine disorders - Other, specify (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Esophageal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Eye disorders - Other, specify (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 4
Facial pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 3 | 3 | 10 | 7 | 14 | 13 | 21
Fever (General disorders) | 2 | 2 | 0 | 2 | 1 | 1 | 3 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 0
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 1 | 4 | 2 | 5
Headache (Nervous system disorders) | 1 | 1 | 0 | 2 | 0 | 7 | 2 | 7
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 2
Heart failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hematuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 4 | 0 | 5
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hot flashes (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 7 | 7 | 6 | 11 | 11
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2
Hypertension (Vascular disorders) | 0 | 2 | 3 | 4 | 2 | 5 | 4 | 10
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 2 | 4 | 2 | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 2
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 2 | 2 | 4 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 4
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 3 | 1 | 14 | 2 | 16
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
INR increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 0 | 3 | 0 | 1 | 1 | 3
Investigations - Other, specify (Investigations) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Localized edema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Lung infection (Infections and infestations) | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 0
Lymphedema (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 2 | 2 | 2 | 1 | 2 | 2 | 5
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 2 | 1 | 3 | 6 | 12 | 9 | 13
Nervous system disorders - Other, specify (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 3
Oral hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 2
Pain (General disorders) | 1 | 1 | 1 | 4 | 2 | 7 | 3 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Platelet count decreased (Investigations) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 3 | 1 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2 | 3 | 6 | 2 | 10 | 6 | 15
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 3 | 0 | 1 | 2 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1 | 5 | 1 | 6
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 2 | 1 | 1 | 2 | 2
Scalp pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Stoma site infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Thromboembolic event (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 2
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 2 | 2 | 3 | 3
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Tremor (Nervous system disorders) | 2 | 1 | 2 | 2 | 2 | 2 | 5 | 3
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Upper respiratory infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
Urinary frequency (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 3
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Vascular disorders - Other, specify (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 3 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 3 | 4 | 3 | 5
Weight loss (Investigations) | 3 | 3 | 0 | 7 | 4 | 8 | 8 | 11
White blood cell decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-31): https://cdn.clinicaltrials.gov/large-docs/63/NCT02244463/Prot_SAP_000.pdf